CLINICAL TRIAL: NCT05633693
Title: Impact of Postural Sway on Cardiovascular Control in Pediatric Patients With Syncope
Brief Title: Postural Sway and Counterpressure Maneuvers for Pediatric Syncope
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); University of British Columbia (Other); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Dr. Victoria Claydon, Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H22-02694
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance
MeSH Terms: conditions — Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counterpressure Maneuvers (Experimental): Counterpressure maneuver (CPM) trials will be performed in front of a neutral wall in silence to ensure that visual or auditory stimuli do not affect movement.
  CPM:
  * Leg crossing and muscle tensing: Legs are crossed while upright and lower body musculature is isometrically contracted (clinical)
  * Crouching: Participant crouches down resting weight on the balls of their feet, pressing calves against the back surface of the thighs (clinical)
  * Exaggerated anterior-posterior sway: Participant sways back and forth with feet planted on ground at a pace/amplitude that is comfortable (discrete)
  * Gluteal clenching: Participant rhythmically tenses and relaxes the gluteal muscles at a pace/duration that is comfortable (discrete)
  Participants serve as their own controls and complete both testing arms.
  Interventions: Behavioral: Counterpressure Maneuvers; Behavioral: Baseline Stand
- Baseline Stand (Sham Comparator): Participants will perform a sit-stand test, followed by 5-minutes of baseline (quiet) standing trial on a force platform while cardiorespiratory responses are recorded.
  Sit-stand test: following 5-minutes of supine rest, the participant will be passively moved into the seated position. They will then be asked to actively move into the standing position.
  Baseline stand: immediately following the sit-stand test, the baseline trial will begin. Participants will stand quietly on the force platform for 5-minutes. This trial will be performed in front of a neutral wall in silence to ensure that visual or auditory stimuli do not affect their movement.
  Participants serve as their own controls and complete both testing arms.
  Interventions: Behavioral: Counterpressure Maneuvers; Behavioral: Baseline Stand

INTERVENTIONS:
Behavioral: Counterpressure Maneuvers — Movements that can aid in delaying or preventing syncope by recruiting skeletal muscle pumping (via compression of major veins by contracting muscle to eject blood through cardiovascular circuit) and increased sympathetic drive (via sustaining an isometric muscle contraction). In this trial, we will be evaluating two clinically recommended isometric maneuvers (crouching, and leg crossing with muscle tensing) and two novel dynamic maneuvers that comprise discrete movement that the investigators have identified in prior work (exaggerated anterior-posterior postural sway, rhythmic gluteal clenching).
  Other Names: Physical counter maneuvers, counter maneuvers,
Behavioral: Baseline Stand — Participants will stand quietly for 5-minutes on a force platform to allow the investigators to assess their typical response to orthostasis.
  Other Names: Quiet standing

SUMMARY:
The investigators are interested in whether discrete counterpressure maneuvers, or muscle movements in the lower body, will boost blood pressure and cardiovascular control in children who faint. We will record cardiovascular responses to maneuvers of exaggerated sway, leg crossing, crouching, and gluteal muscle tensing in children who faint (N=20), as well as their height, weight, muscularity, and pubertal (Tanner) stage. Autonomic cardiovascular control will be measured using a Valsalva manoeuvre (expiration against a closed airway for 20 seconds) and a supine-stand test. The primary outcomes are noninvasive measures of cardiovascular responses to the maneuvers (blood pressure, cerebral blood flow, and stroke volume (volume of blood pumped per heartbeat). Comparisons will be made across levels of sex, diagnosis, Tanner stage, muscularity, height, and degree of autonomic control.

DETAILED DESCRIPTION:
Purpose: The primary purpose of this investigation is to determine whether discrete counterpressure maneuvers (CPM; exaggerated sway, rhythmic gluteal muscle clenching) can demonstrably improve the return of blood to the heart and the blood pressure in paediatric patients with recurrent uncomplicated syncope (fainting), and to assess whether these discrete CPM are more effective than those commonly recommended in the clinic (leg crossing, crouching).

Protocol: Volunteers (n=35) will be asked to attend one testing session. Testing will take approximately 1.5 hours. Tests will usually be conducted in the mornings. On the day of the test volunteers will be asked to have only a light breakfast avoiding caffeine, and should avoid strenuous exercise for at least 12 hours prior to testing. Female participants that have reached menarche will be asked to make a note of the date of their last period (we would prefer to schedule testing on a day when they do not have, or expect, their period because this may influence orthostatic tolerance).

Prior to testing volunteers will be asked a brief narrative medical history including questions regarding their syncopal diagnosis, and as to whether they have any known cardiovascular or neurological disease, are taking any medications, and questions about general cardiovascular risk factors such as smoking, and alcohol consumption. Participants will also be asked to complete a short questionnaire about their fainting spells. All participants will be asked to self-identify their stage in pubertal development ("Tanner" stage) based on drawn images of biologically male and female bodies at each stage. If participants to not identify with these images, have difficulty answering the question, or do not wish to answer for any reason, they do not have to do so (and are not required to provide this reason). Participants will then complete the PEDS-QL (Pediatric Quality of Life Inventory) and PAQ (Physical Activity Questionnaire). Measures of height, weight and muscle mass will be taken using a height chart and impedance-based weighing scale. Anthropometric measurements of body composition (skinfold thickness: bicep, tricep, thigh, medial calf; circumference: mid-upper arm, mid-thigh, mid-calf) will also be performed. A copy of the prompt sheet used by the investigators to facilitate taking the medical history is included with the submission. This form outlines the medical history data collected in general terms and is used to guide a narrative history. Participants will be asked to empty their bladder in the nearby washroom, and to retain a sample of their urine for testing for sodium levels (a marker of salt intake and hydration). One the urine has been tested it will be discarded. No biological samples will be retained. A brief instruction on the different tests of nervous system function ("Valsalva maneuver") and movement patterns (see below) will occur.

Participants will then be asked to lie down on a standard hospital style examination bed. The investigators will then attach the following CSA approved cardiovascular monitoring (all monitors are non-invasive and painless):

1. A standard 3 lead electrocardiogram (ECG) will be recorded to assess heart rate and rhythm.
2. Beat-to-beat blood pressure will be determined using the Finometer blood pressure monitoring device. This consists of a small Velcro cuff placed around the middle finger that pulses gently against the digital arteries and records and displays blood pressure with every heartbeat.
3. End tidal gases will be sampled using a nasal cannula. This is to enable us to evaluate any influence of possible hyperventilation and the associated decreases in carbon dioxide on cerebral blood flow.
4. Cerebral blood flow will be determined in the middle cerebral artery using Doppler ultrasound. An ultrasound probe will positioned on the skin overlying the temple and held in place with a head band. Participants can move their head freely when wearing the ultrasound probe.
5. Brachial blood flow will be determined using an ultrasound probe positioned overlaying the brachial artery in the upper arm. The probe will be positioned on the participant's arm using an adjustable holder. It will only be in place during the initial supine period, and the Valsalva maneuver.

Once the monitors are in place, participants will be asked to perform two Valsalva manoeuvres, which is a test of parasympathetic and sympathetic control of the circulatory system and cardiac baroreflex function. During this test, participants will blow out against a closed tube to produce a Valsalva strain (performed as though they were blowing up a balloon that would not inflate, generating a pressure of 40mmHg) and sustain this for 20 seconds. The tube will be connected to a manometer (provides a pressure reading) so the participant can regulate their expiratory pressure. The participant will perform one Valsalva maneuver while lying supine, and a second while sitting upright. Responses will be monitored continuously using the equipment mentioned above.

Next, the participants will complete a 5-minute supine rest period, after which they will be asked to rise from the supine to the standing position and stand on the force platform while we record their cardiovascular and cerebrovascular responses for 5 minutes. Volunteers will stand without shoes, and will be asked not to move their feet for the duration of each standing trial. Following this, volunteers will perform four more bouts of a 5-minute supine period, followed by a 5-minute standing period on the force platform. During each of these trials, they will perform one of the following movements:

1. Exaggerated anterior-posterior sway: rocking the body in a fore-aft motion, as far as comfortably possible without raising the heels or toes off the force platform
2. Gluteal clenching: rhythmic tensing of the thighs and buttocks
3. Crouching: lowering body to the floor in a crouched position
4. Leg crossing with muscle tensing: standing with legs crossed for the first 4 minutes of the trial, clenching legs in the crossed position for the final minute.

These standing trials will be completed in a randomized order. Following their completion, testing will be concluded. The monitoring equipment will be removed and any residue from the ultrasound gel will be wiped away by the participant.

Testing will stop if the volunteer experiences symptoms of presyncope, decreased blood pressure (<80mmHg systolic pressure for greater than 5 consecutive heart beats), slowing of the heart rate (new onset bradycardia below 50bpm), or at the participant's request. In such an instance the participant will be asked to lie flat until any symptoms or signs of presyncope resolve. If participants meet criteria to stop testing during one of the standing phases, but haven't yet finished all standing phases, they can decide if they want to try the next standing phase, or stop testing all together.

ELIGIBILITY:
Inclusion Criteria:

We are looking for English speaking pediatric patients aged 6-18 years with a diagnosis of recurrent fainting (at least two episodes of fainting with loss of consciousness or near loss of consciousness in the last year) of a vasovagal origin or associated with the postural orthostatic tachycardia syndrome (POTS) (as determined by a paediatric cardiologist) to take part in this study.

Exclusion Criteria:

Those with a diagnosis of recurrent fainting accompanied by any of the following will not be eligible to take part:

Known history of:

* Suspected or confirmed cardiac arrhythmia (e.g., Wolff-Parkinson-White, Long QT)
* Traumatic head injury
* New presentation of a seizure disorder OR epilepsy recurrence
* Overdose or intoxication
* Structural heart disease
* Cardiovascular disease including hypertension, diabetes, or renal disease
* Hypoglycemia
* Physical and/or psychological disability that impact their ability to complete the tests

Female participants of childbearing age will be excluded if they are pregnant, or think they might be. Participants who are taking any cardiovascular acting medications, including treatment for cardiovascular disease, or medications for orthostatic syncope (e.g. fludrocortisone, slow-release sodium chloride, β-blockers, midodrine) will be excluded from the study.

In order to reduce the likelihood of transmission of COVID-19, participants will only be eligible to participate in the study if they have received full immunisation against COVID-19 according to current Health Canada guidelines. Accordingly, participants will be asked to provide evidence of their vaccination status in order to take part in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Relationship between postural movement and stroke volume | Final minute of maneuver performance
  We will correlate these two parameters using both time and frequency domain approaches. We will compare this between the five movement conditions using a one-way repeated measures ANOVA.

SECONDARY OUTCOMES:
Relationship between anthropometry and response magnitude | Final minute of maneuver performance
  We will evaluate the relationship between responses to the CPM and factors of muscle mass and height. We will evaluate this using correlation, regression, and AIC analyses.
Relationship between tanner stage and response magnitude | Final minute of maneuver performance
  We will compare responses across tanner stages using a 2-way repeated measures ANOVA. We will also consider sex differences in cardiovascular responses to the maneuver, again using a 2-way repeated measures ANOVA
Relationship between autonomic control and response magnitude | Final minute of maneuver performance, response to maneuver release.
  We will use responses to the Valsalva maneuver and sit-stand test to determine participant autonomic control. Relationships between autonomic control will be evaluated using correlation/regression/AIC analyses. Comparisons between syncopal diagnoses will be made using a 2-way Repeated Measures ANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Claydon, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke DA, Medow MS, Taneja I, Ocon AJ, Stewart JM. Initial orthostatic hypotension in the young is attenuated by static handgrip. J Pediatr. 2010 Jun;156(6):1019-1022.e1. doi: 10.1016/j.jpeds.2010.01.035. Epub 2010 Mar 28. PMID 20350727
- [Background] Williams EL, Khan FM, Claydon VE. Counter pressure maneuvers for syncope prevention: A semi-systematic review and meta-analysis. Front Cardiovasc Med. 2022 Oct 13;9:1016420. doi: 10.3389/fcvm.2022.1016420. eCollection 2022. PMID 36312294
- [Background] Inamura K, Mano T, Iwase S, Amagishi Y, Inamura S. One-minute wave in body fluid volume change enhanced by postural sway during upright standing. J Appl Physiol (1985). 1996 Jul;81(1):459-69. doi: 10.1152/jappl.1996.81.1.459. PMID 8828698
- [Background] Claydon VE, Hainsworth R. Increased postural sway in control subjects with poor orthostatic tolerance. J Am Coll Cardiol. 2005 Oct 4;46(7):1309-13. doi: 10.1016/j.jacc.2005.07.011. PMID 16198849
- [Background] Stewart JM, Medow MS, Montgomery LD, McLeod K. Decreased skeletal muscle pump activity in patients with postural tachycardia syndrome and low peripheral blood flow. Am J Physiol Heart Circ Physiol. 2004 Mar;286(3):H1216-22. doi: 10.1152/ajpheart.00738.2003. Epub 2003 Oct 23. PMID 14576081
- [Background] Claydon VE, Hainsworth R. Postural sway in patients with syncope and poor orthostatic tolerance. Heart. 2006 Nov;92(11):1688-9. doi: 10.1136/hrt.2005.083907. No abstract available. PMID 17041121
- [Background] van Dijk N, Quartieri F, Blanc JJ, Garcia-Civera R, Brignole M, Moya A, Wieling W; PC-Trial Investigators. Effectiveness of physical counterpressure maneuvers in preventing vasovagal syncope: the Physical Counterpressure Manoeuvres Trial (PC-Trial). J Am Coll Cardiol. 2006 Oct 17;48(8):1652-7. doi: 10.1016/j.jacc.2006.06.059. Epub 2006 Sep 26. PMID 17045903
- [Background] Coupal KE, Heeney ND, Hockin BCD, Ronsley R, Armstrong K, Sanatani S, Claydon VE. Pubertal Hormonal Changes and the Autonomic Nervous System: Potential Role in Pediatric Orthostatic Intolerance. Front Neurosci. 2019 Nov 12;13:1197. doi: 10.3389/fnins.2019.01197. eCollection 2019. PMID 31798399